CLINICAL TRIAL: NCT02358096
Title: A Phase 2, Double-Blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of ASP8232 as Add-On Therapy to Angiotensin Converting Enzyme Inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) in Reducing Albuminuria in Patients With Type 2 Diabetes and Chronic Kidney Disease
Brief Title: A Study to Evaluate ASP8232 as Add-On Therapy to Angiotensin Converting Enzyme Inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) in Reducing Albuminuria in Patients With Type 2 Diabetes and Chronic Kidney Disease
Acronym: ALBUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8232-CL-0004; 2014-002349-23 (EudraCT Number)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes
Keywords: Chronic Kidney Disease; Type 2 Diabetes; ASP8232
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — ASP8232

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP8232 (Experimental): ASP8232 administered once daily
  Interventions: Drug: ASP8232
- Placebo (Placebo Comparator): Placebo administered once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8232 — oral capsule
  Arms: ASP8232
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of ASP8232 in reducing Urinary Albumin to Creatinine Ratio (UACR) in subjects with Type 2 Diabetes Mellitus (T2DM) and Chronic Kidney Disease (CKD) at 12 weeks compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have an estimated glomerular filtration rate (eGFR) ) >=25 and <75 ml/min/1.73m2.
* Subject must have a documented diagnosis of T2DM and received anti-diabetic medication (oral and/or parenteral) for at least 1 year prior to screening
* Subject's glycated hemoglobin (HbA1c) level is < 11.0% (<97 mmol/mol) at screening.
* Subject is on a stable therapy with an angiotensin-converting-enzyme (ACE) inhibitor or angiotensin receptor blockers (ARB) for at least 3 months prior to screening.
* Subject who receives anti-hypertensive treatment, non-insulin anti-diabetic agents and/or vitamin D receptor activators at screening needs to be on stable therapy for at least 3 months prior to screening. Subjects on insulin therapy may have the insulin type/dose/schedule adjusted even during the 3 months prior to screening.
* If the subject has been subjected to specific dietary interventions then this has to be stable over the past 3 months prior to screening visit.
* Subject's UACR is ≥ 200 and ≤ 3000 mg/g in a first morning void (FMV) sample at screening AND the geometric mean UACR of all FMV samples at visit 4 and at visit 5 is ≥ 200 and ≤ 3000 mg/g AND the UACR in at least 3 FMV samples at visit 4 and visit 5 is ≥ 200 mg/g.

Exclusion Criteria:

* Subject is on, or previously received, renal replacement therapy (e.g. dialysis or kidney transplantation).
* Subject has obstructive uropathy or other causes of renal impairment not related to parenchymal renal disorder and/or disease of the kidney; or subject currently has or has had in the past renal disease secondary to malignancy.
* Subject's renal impairment and/or albuminuria is considered to be of other origin than Diabetic Kidney Disease.
* Subject has known (auto-) immune disorder and/or received immunosuppression for more than 2 weeks, cumulatively, within 12 weeks prior to screening or anticipated need for immuno-suppressive therapy during the study.
* Subject has active urinary tract infection which requires treatment or clinically significant infection at the time of screening or randomization
* Subject is diagnosed with type 1 diabetes mellitus or diabetes mellitus with unclear etiology.
* Subject has a sitting systolic blood pressure (SBP) <90 or >160 mmHg and/or a diastolic blood pressure (DBP) >90 mmHg at screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Mean change of log transformed urinary albumin to creatinine ratio (UACR) from baseline to end of treatment | Baseline and end of treatment (12 weeks)

SECONDARY OUTCOMES:
Proportion of subjects with either >30% or >40% or >50% reduction in UACR from baseline to end of treatment | Baseline and end of treatment (12 weeks)
Mean change of log transformed albumin excretion rate (AER) from baseline to end of treatment | Baseline and end of treatment (12 weeks)
Proportion of subjects with either >30% or >40% or >50% reduction in AER from baseline to end of treatment | Baseline and end of treatment (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma Europe B.V.
Locations (57):
- Czechia (5):
  - Site CZ42002, Brno
  - Site CZ42003, České Budějovice
  - Site CZ42005, Prague
  - Site CZ42001, Prague
  - Site CZ42004, Prague
- Denmark (6):
  - Site DK45016, Copenhagen
  - Site DK45004, Gentofte Municipality
  - Site DK45001, Herlev
  - Site DK45002, Hillerød
  - Site DK45007, Holsterbro
  - Site DK45006, Viborg
- Germany (4):
  - Site DE49004, Berlin
  - Site DE49002, Düsseldorf
  - Site DE49008, Elsterwerda
  - Site DE49003, Heidelberg
- Hungary (9):
  - Site HU36002, Balatonfüred
  - Site HU36016, Budapest
  - Site HU36010, Budapest
  - Site HU36003, Hatvan
  - Site HU36012, Kaposvár
  - Site HU36017, Székesfehérvár
  - Site HU36007, Szigetvár
  - Site HU36005, Szikszó
  - Site HU36018, Veszprém
- Italy (5):
  - Site IT39007, Bergamo
  - Site IT39005, Pavia
  - Site IT39002, Piacenza
  - Site IT39012, Rome
  - Site IT39004, Turin
- Netherlands (3):
  - Site NL31004, Rotterdam, South Holland
  - Site NL31001, Dordrecht
  - Site NL31003, Hoogeveen
- Poland (11):
  - Site PL48026, Lodz
  - Site PL48008, Lodz
  - Site PL48004, Lodz
  - Site PL48027, Oświęcim
  - Site PL48001, Poznan
  - Site PL48003, Płock
  - Site PL48022, Radom
  - Site PL48006, Rzeszów
  - Site PL48005, Sopot
  - Site PL48002, Torun
  - Site PL48025, Warsaw
- Spain (10):
  - Site ES34001, Barcelona
  - Site ES34005, Barcelona
  - Site ES34004, Barcelona
  - Site ES34002, Barcelona
  - Site ES34007, Ciudad Real
  - Site ES34006, Lugo
  - Site ES34008, Madrid
  - Site ES34012, Madrid
  - Site ES34010, Majadahonda
  - Site ES34003, Palma de Mallorca
- United Kingdom (4):
  - Site GB44004, Burton-on-Trent
  - Site GB44001, Chester
  - Site GB44005, London
  - Site GB44003, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] de Zeeuw D, Renfurm RW, Bakris G, Rossing P, Perkovic V, Hou FF, Nangaku M, Sharma K, Heerspink HJL, Garcia-Hernandez A, Larsson TE. Efficacy of a novel inhibitor of vascular adhesion protein-1 in reducing albuminuria in patients with diabetic kidney disease (ALBUM): a randomised, placebo-controlled, phase 2 trial. Lancet Diabetes Endocrinol. 2018 Dec;6(12):925-933. doi: 10.1016/S2213-8587(18)30289-4. Epub 2018 Nov 6. PMID 30413396
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=266